CLINICAL TRIAL: NCT07194382
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Proof of Concept (POC) Study Evaluating the Safety, Tolerability, and Efficacy of Nintedanib Solution for Inhalation (AP02) in Participants With Idiopathic Pulmonary Fibrosis (IPF) (AURA-IPF)
Brief Title: AURA-IPF: A Randomized Phase 2 Study to Evaluate the Safety and Efficacy of AP02 (Nintedanib Solution) in IPF
Acronym: AURA-IPF
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Avalyn Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP02-003
Record Dates: First submitted 2025-09-04; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Idiopathic Pulmonary Fibrosis; IPF; AP02
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo BID (Placebo Comparator): Placebo solution for Inhalation
  Interventions: Drug: Placebo
- AP02 low dose BID (Active Comparator): Nintedanib solution for Inhalation
  Interventions: Drug: AP02
- AP02 high dose BID (Active Comparator): Nintedanib solution for Inhalation
  Interventions: Drug: AP02

INTERVENTIONS:
Drug: AP02 — Oral inhalation solution
  Arms: AP02 high dose BID; AP02 low dose BID
Drug: Placebo — Placebo oral inhalation solution
  Arms: Placebo BID

SUMMARY:
This study will evaluate the impact Nintedanib Solution for Inhalation (AP02) has on lung function and key measures of fibrosis in adult patients with idiopathic pulmonary fibrosis (IPF) as well as assess its safety and tolerability.

Adults 40 years of age or older with IPF who meet the inclusion and exclusion criteria can participate in this study if they are not currently on treatment for IPF, and if treated with oral nintedanib or pirfenidone, have stopped the medication for at least 3 months.

Researchers will compare two different doses of AP02 to a placebo (a look-alike substance that contains no drug) to see if AP02 works to treat IPF. Participants are put into 1 of 3 groups randomly, which means by chance and will take AP02 or a placebo two times every day for 12 weeks by using a nebulizer, which is a device that provides medicine to the lungs via inhalation.

Participants will visit the office 6 times and receive 1 phone call over a 16-week period. At site visits doctors regularly perform breathing tests that measure how well the lungs are working, give the patient questionnaires and will check the participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥40 years at the time of signing the written informed consent form
* Diagnosis of idiopathic pulmonary fibrosis (IPF) as defined by American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/ Asociación Latinoamericana de Tórax IPF guidelines within 5 years
* Combination of High-Resolution Computerized Tomography (HRCT) pattern, and if available, surgical lung biopsy pattern consistent with diagnosis of IPF
* In a stable condition and suitable for study participation based on the results of medical history, physical examination, vital signs, 12-lead ECG, and laboratory evaluation
* Forced vital capacity (FVC) ≥45% predicted of normal
* Lung diffusion test (DLCO) corrected for hemoglobin (Hgb) ≥30% and ≤80% predicted of normal.
* Women and men of childbearing potential must use highly effective contraception measures until 90 days after the last dose of study drug.

Exclusion Criteria:

* Current treatment with oral nintedanib, oral pirfenidone, or previous treatment with oral nintedanib or oral pirfenidone within 3 months prior to screening. Participants who have taken both oral nintedanib and pirfenidone together as a treatment will not be able to join the study.
* Forced expiratory volume (FEV) in the first second/FVC (FEV1/FVC) ratio ≥0.7 based on pre-bronchodilator value
* Participants with a history of serious cardiovascular disease, bleeding problems or significant liver or kidney disease (as defined in the study protocol)
* History of diverticular disease or abdominal surgery within 4 weeks prior to screening visit
* History of cancer within the past 5 years (except for certain types explained in the protocol)
* Participants who have smoked within the past 3 months prior to screening, who are not willing to stop smoking during the study, or who currently use illegal drugs or drugs of abuse
* Female participants who are pregnant or nursing
* Use of any investigational drugs including those for IPF within the past 30 days prior to screening

Further inclusion/exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the morning pre-dose forced vital capacity at Week 12 | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
Time to disease progression | From enrollment to the end of treatment at 12 weeks
  Disease progression is defined as forced vital capacity (FVC) percent predicted decline of ≥10% prior to Week 12, respiratory hospitalization, or death.
To evaluate the change from baseline in quantitative lung fibrosis score | From enrollment to the end of treatment at 12 weeks
  Change in lung fibrosis score.